CLINICAL TRIAL: NCT01350700
Title: Scar Formation and Quality of Life Assessment in Subjects (Adults & Children) Following Treatment With Debrase Compared to Standard of Care (SOC)
Brief Title: Long Term Follow up of Scars Formation and Quality of Life Assessment Study
Status: Completed | Type: Observational
Sponsor: MediWound Ltd (Industry)
Responsible Party: Dina Kofler ,Clinical Project Manager, MediWound Ltd, Bio-technology company, MediWound Ltd
Other Study IDs: MW2012-01-02
Record Dates: First submitted 2011-05-08; First posted 2011-05-10 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2011-05

CONDITIONS: Scars Formation; Quality of Life
Keywords: QOL
MeSH Terms: interventions — Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients that were treated in MW2004-011-02 study with Debrase
  Interventions: Other: Scars assessment & QOL
- Patients that were treated in MW2004-011-02 with SOC
  Interventions: Other: Scars assessment & QOL

INTERVENTIONS:
Other: Scars assessment & QOL — Scar assessment and quality of life questionnaires

SUMMARY:
In previous study (MW2004-011-02), patients with burn wounds had their damaged skin removed by either standard of care treatment or by Debrase Gel Dressing (DGD), which is composed of enzymes that dissolve the damaged skin selectively (DGD removes only the damaged skin and not other parts of the skin).

The burn wound, like any other wound, heals by the formation of scar at the injured site in order to replace the destroyed tissues. Scarring is not a static process, but rather a dynamic one, changing over time, especially during the first 24 months post-injury.

Scars and patients' quality of life from two treatment arms (DGD and SOC) will be compared in order to evaluate the long term influence of damaged skin removal and wound care techniques on scar formation and maturation.

ELIGIBILITY:
Inclusion criteria

1. Adults and children who had participated and completed study MW2004-11-02.
2. Subjects must be willing and able to sign a written informed consent prior to study entry (by subject or by a guardian, when applicable).

Ages: 4 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients that have previously participated in MW2004-011-02 study
Sampling Method: Non-Probability Sample
Enrollment: 148 (Estimated)
Dates: Start 2011-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11-22 (Actual)

PRIMARY OUTCOMES:
1. Scar assessment of target wounds that have been treated by Debrase or SOC during MW2004-11-02 using Modified Vancouver Scar Scale (MVSS) | Approximately 2 years after wound closure
  Assesment of scars will be done using the Modified Vancouver Scar Scale
2. To evaluate and compare the Quality of Life (QoL) in adult and children that their burn wounds were treated with Debrase or SOC in study MW2004-11-02 | Approximately 2 years after wound closure
  2. A Quality of Life (QoL) assessment will be performed in burn victims using a Short Form 36 (SF-36) and Burn Outcomes Questionnaire (BOQ).

CONTACTS AND LOCATIONS:
Overall Officials: Jan Koller, MD,PhD, Principal Investigator — Department Head of Burs and Reconstructive Surgery
Locations (1):
- Clinic of Burns and reconstructive surgery hospital, Košice, Slovakia